CLINICAL TRIAL: NCT01381952
Title: XRES4 Neuro Claim Study
Brief Title: Image Quality and Radiation Dose in Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Philips Medical Systems (Industry)
Responsible Party: Principal Investigator, Michael Söderman, MD, PhD, Karolinska University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: KUH-PMS-01
Record Dates: First submitted 2011-06-20; First posted 2011-06-27 (Estimated); Results first posted 2014-05-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-04

CONDITIONS: Arteriovenous Malformations; Aneurysm; Stenosis; Dural Arteriovenous Malformations
Keywords: X-ray; Image processing; Neuro angiography; Radiation exposure
MeSH Terms: conditions — Arteriovenous Malformations; Aneurysm; Constriction, Pathologic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reduced radiation dose (ClarityIQ) (Experimental): Low dose DSA (75% reduction compared to normal dose) with novel X-ray imaging technology
  Interventions: Radiation: Low dose DSA (75% reduction compared to normal dose) with novel X-ray imaging technology.
- Normal radiation dose (AlluraXper) (Active Comparator): Normal dose DSA with conventional X-ray technology.
  Interventions: Radiation: Normal dose DSA with conventional X-ray technology

INTERVENTIONS:
Radiation: Low dose DSA (75% reduction compared to normal dose) with novel X-ray imaging technology. — Digital substraction angiography (DSA) with reduced dose settings (75% reduction expected) in combination with conventional X-ray imaging technology.
  Other Names: ClarityIQ
  Arms: Reduced radiation dose (ClarityIQ)
Radiation: Normal dose DSA with conventional X-ray technology — Digital substraction angiography (DSA) with normal dose settings in combination with conventional X-ray imaging technology.
  Other Names: AlluraXper
  Arms: Normal radiation dose (AlluraXper)

SUMMARY:
ClarityIQ is a novel X-ray imaging technology, that combines advanced real-time image noise reduction algorithms, with state-of-the-art hardware to reduce patient entrance dose significantly. This is realized by anatomy-specific optimization of the full acquisition chain (grid switch, beam filtering, pulse width, spot size, detector and image processing engine) for every clinical task individually. Furthermore, smaller focal spot sizes and shorter pulses are used, which are known to positively influence image quality . The final effect on the clinical image quality is investigated in this study.

DETAILED DESCRIPTION:
The advent of interventional neuroradiology (INR) has changed the treatment of neurovascular diseases by reducing the procedural invasiveness and the recovery time needed by patients, thus improving clinical outcome. However, INR procedures often require many high-quality digital substraction angiography (DSA) runs and long total fluoroscopy times, which can result in patients being exposed to considerable radiation doses levels.

In order to introduce a dose reduction technology the most important aspect is to validate the diagnostic image information. Philips has developed a real-time noise reduction algorithm for DSA in neuroradiology that is capable to reduce the patient entrance dose by 75% without loss of image quality.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Normal kidney function
* Neurologically intact
* Planned for diagnostic angiography or endovascular treatment

Exclusion Criteria:

* Pregnancy
* Other conditions that limit the use of contrast media or ionizing radiation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Söderman, MD, PhD, Principal Investigator — Karolinska University Hospital; Tommy Andersson, MD, PhD, Principal Investigator — Karolinska University Hospital; Staffan Holmin, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Solna, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment of patients occurred between 22 June 2011 and 11 August 2011
Pre-assignment Details: 20 patients enrolled the study; 16 patients were undergoing diagnostic neuroangiography and 4 were undergoing INR procedures for different pathological conditions. All signed patient consent.
Groups:
- AlluraXper - ClarityIQ: Angiogram with AlluraXper subsequently followed by angiogram with ClarityIQ
Period: Overall Study
Arm/Group | AlluraXper - ClarityIQ
Started | 20
Collected Dose and Image Information | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- AlluraXper - ClarityIQ: Angiogram with AlluraXper followed by angiogram with ClarityIQ
Arm/Group | AlluraXper - ClarityIQ
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Number; unit: participants]
  Sweden | 20

OUTCOME MEASURES:

1. Primary Outcome: Image Quality. For Each Included Participant 2 Images (1 AlluraXper; 1 AlluraClarity) Were Evaluated.
Description: The images were evaluated in randomized, blinded, offline readings. The anonymized images were displayed in pairs, i.e. the reference image run on one monitor (randomly left or right side) with the corresponding quarter-dose image run on the adjacent monitor. Three neuroradiologists graded the arterial, capillary, and venous phases separately. For each characteristic the images quality (IQ) were rated on a scale of 1 to 5 as 1 (very poor), 2 (mediocre), 3 (average), 4 (good), 5 (very good/excellent). An overall IQ score (3-15) was calculated as the sum of the score for these characteristics.
  A paired Student's t test is used to compare the overall IQ score between the 2 imaging techniques. If the upper limit of the 97.5% one-sided CI for the difference overall IQ between the two treatment groups does not exceed the pre-defined non-inferiority margin of 2.5 Clarity will be declared non-inferior to the current image acquisition settings for DSA.
Time Frame: 1 day
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- AlluraXper; Allura Clarity: Angiogram with AlluraXper followed by angiogram with ClarityIQ
Arm/Group | AlluraXper | Allura Clarity
Number analyzed (Participants) | 20 | 20
Scores on a scale
  Investigator 1 | 9.4 [8.99 to 9.81] | 11.9 [11.33 to 12.42]
  Investigator 2 | 13.1 [12.75 to 13.45] | 14.1 [13.75 to 14.42]
  Investigator 3 | 11.1 [10.59 to 11.66] | 12.1 [11.42 to 12.68]

2. Secondary Outcome: Radiation Dose Measurements: Dose Area Product (DAP)
Description: Percentage of dose reduction of ClarityIQ vs. AlluraXper in Dose Area Product (DAP) calculated by DAP/frame.
Time Frame: Participants were followed for the duration of the procedure
Population: All patients with recorded dose information and images for both angiograms were included (n=20)
Measure: Mean (Standard Deviation); unit: percentage of dose reduction
Arm/Group | AlluraXper - ClarityIQ
Number analyzed (Participants) | 20
percentage of dose reduction | 72.4 (1.95) [71.5 to 73.3]

3. Other Pre Specified Outcome: Radiation Dose Measurements: Air Kerma (AK)
Description: Percentage of dose reduction of ClarityIQ vs. AlluraXper in Air Kerma (AK) calculated by AK/frame.
Time Frame: Participants were followed for the duration of the procedure
Population: All patients with recorded dose information and images for both angiograms were included (n=20)
Measure: Mean (Standard Deviation); unit: percentage of dose reduction
Arm/Group | AlluraXper - ClarityIQ
Number analyzed (Participants) | 20
percentage of dose reduction | 74.6 (0.9)

ADVERSE EVENTS:
Arm/Group | AlluraXper - ClarityIQ
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less